CLINICAL TRIAL: NCT06160245
Title: Effect of Core Stabilization Exercises on Cervical Sagittal Balance Parameters in Forward Head Posture
Brief Title: Core Stabilization Exercises in Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Mohamed Shabana, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSEs in FHP
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Forward Head Posture
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stability exercise (Experimental): This group will receive core stabilization exercises ( MCGILL 2008), in addition to postural correction exercises described by (HARMAN 2005)
  Interventions: Other: exercise therapy
- traditional exercise (Active Comparator): This group will receive only postural correction exercises described by (HARMAN 2005)
  Interventions: Other: exercise therapy

INTERVENTIONS:
Other: exercise therapy — core stabilization exercises

SUMMARY:
Based on the reviewed literature, Core Stabilization Exercises (CSEs) have been shown to have positive effects on patients with low back pain. To our knowledge, very few studies have examined the impact of CSEs on neck pain, particularly in patients with forward head posture (FHP), despite that several authors suggested that FHP may be caused by lumbopelvic malalignment.

Therefore, the purpose of the study is to assess how CSEs may affect the cervical sagittal balance parameters (CSB) in patient with FHP.

DETAILED DESCRIPTION:
After the patient fills the consent form, the Craniovertebral angle will be measured by taking a photograph, then this photograph will be analysed by the KINOVEA software.

If the CVA is less than 50 degrees, he/she will have a lateral x-ray on the cervical spine to measure the radiographic variables of the CSB parameters. These variables will be assessed and quantified by Image J software.

The patients will be classified randomly into 2 groups, the intervention and control groups. The intervention will receive CSEs program and Postural Correction Exercises (PCEs) program, but control group will receive only PCEs program.

Both programs will be implemented for 6 weeks 3 times/ week and after 6 weeks, patients will be reassessed again to determine the difference.

ELIGIBILITY:
Inclusion Criteria:

* CVA less than 50 degrees/ neck pain for about 4 weeks

Exclusion Criteria:

* Vertebrobasilar insufficiency/ cervical surgery/ cervical or TMJ fracture

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
cervical sagittal vertical alignment | baseline, week 6
  calculated by measuring the horizontal distance between the posterosuperior corner of the C7 vertebral body and a plumb line drawn from the centroid of C2
T1 slope angle | baseline, week 6
  he angle formed by drawing a line along the superior endplate of T1 and horizontal reference line at the median sagittal cervical vertebra from the CT radiographs
craniovertebral angle | baseline, week 6
  the intersection of a horizontal line passing through the C7 spinous process and a line joining the midpoint of the tragus of the ear to the skin overlying the C7 spinous process.

SECONDARY OUTCOMES:
numerical pain rating scale | baseline, week 6
  patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity [1]. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible
neck disability index | baseline, week 6
  a standard instrument for measuring self-rated disability due to neck pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Cairo University & AXA One-Health clinics Korba branch, Giza, Egypt

REFERENCES:
- [Derived] Shabana AMM, Ashour RS, Yamany AS, Hanafy AF. Radiographic and clinical effects of core stabilization on cervical pain and sagittal balance in forward head posture: a randomized controlled trial. Asian Spine J. 2026 Jan 6. doi: 10.31616/asj.2025.0297. Online ahead of print. PMID 41490718
- [Derived] Shabana AMM, Hanafy AF, Yamany AS, Ashour RS. Effect of core stabilization exercises on cervical sagittal balance parameters in patients with forward head posture: a randomized controlled trial in Egypt. Asian Spine J. 2025 Feb;19(1):85-93. doi: 10.31616/asj.2024.0328. Epub 2025 Jan 20. PMID 39829179